CLINICAL TRIAL: NCT05589506
Title: Rehabilitation of Partial Edentulism Through the Use of Polyetheretherketone (PEEK) Removable Partial Denture (RPD)
Brief Title: Partial Rehabilitation Using a PEEK-acrylic Resin Removable Partial Denture
Acronym: PEEKPilotRPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Invibio Ltd, producer of the PEEK material decided to leave the market and stop production.
Sponsor: Malo Clinic (Other)
Collaborators: Invibio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEEKPilotRPD
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prosthesis Survival
Keywords: prosthesis; removable partial denture; PEEK
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Removable partial denture PEEK (Experimental): Removable partial denture using PEEK-acrylic resin
  Interventions: Device: Removable partial denture PEEK

INTERVENTIONS:
Device: Removable partial denture PEEK — A removable partial denture incorporating PEEK and acrylic resin in its composition used as definitive prosthesis to rehabilitate partial edentulism in the maxilla or mandible.
  Other Names: PEEK prosthesis

SUMMARY:
The goal of this observational study is to evaluate the outcome of a Poly-ether-ether-ketone - acrylic resin removable partial denture used in partial edentulous rehabilitation after one year of follow-up. The main question it aims to answer is:

- What is the survival outcome of partial rehabilitations using Poly-ether-ether-ketone-acrylic resin removable partial dentures? The participants will receive a definitive removable partial denture incorporating Poly-ether-ehter-ketone.

DETAILED DESCRIPTION:
Folowing the recent applications of polyetheretherketone (PEEK) material in Dentistry it is necessary to further extend the evaluation to the use of Removable Partial Denture (RPD) rehabilitations. To test this, the study design to be used will be a single-centre, prospective observational cohort study to evaluate the short term outcome of the Removal Partial Denture (RPO) supported rehabilitations. The sample of this study consists in 10 patients consecutively treated. The cohort will be evaluated at baseline, RPD design, dental fitting, follow-up assessment at 4 weeks, 6 and 12 months after dental loading regarding: JUVORA prosthetic survival including repair and relining, assessment of the adaptation of the RPD frame, adaptation of the tissue base areas and their relationship to the frame adaptation, functional evaluation, aesthetics assessment (staining, color stability, anatomic form), oral health assessment of the RPD abutment teeth periodontium (plaque index, gingival index, probing pocket depths, bleeding on probing, mobility) incidence of mechanical complications (loosening or fracture of prosthetic components), patient assessment of RPD comfort, aesthetics and chewing ability; assessment of RPD preparation (technician satisfaction) concerning laboratory preparation time, clinical operative time and costs.

ELIGIBILITY:
Inclusion Criteria:

* partial edentulism with at least a posterior natural tooth occlusaI stop (molar or premolar), defined as Kennedy's Class I, Class lI or Class lII,
* occlusal spacing (static and dynamic) around clasp assembly including the occlusal rest;
* previous denture wearing experience,
* stable oral health in terms of absence of disease activity affecting the periodontium, caries, pulp and the structural/aesthetic integrity of restored teeth.
* Subjects who, in the opinion of the Investigator, are able to understand this clinical study, co-operate with the procedures and are willing to return to the clinic for all the required post-operative follow-ups.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained.

Exclusion Criteria:

* Female Subjects who are pregnant;
* Subjects requiring extensive treatment prior to the provision of a removable partial denture;
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-ups or treatment outcomes;
* Subjects who are currently enrolled in a clinical study;
* Subjects requiring or currently having ongoing orthodontic treatment;
* Subjects with an opposing Removable Partial Denture (RPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Survival of the prosthesis | one year
  Evaluation of the survival for the PEEK-acrylic resin removable partial denture; nominal (survival,failure)

SECONDARY OUTCOMES:
Assessment of the adaptation of the RPD frame | one year
  Nominal: 0: adapted; 1: not adapted
Function of RPD is excellent | one year
  5-point Likert scale: strongly agree, agree, neutral, disagree, strongly disagree
Aesthetics of RPD are excellent | one year
  5-point Likert scale: strongly agree, agree, neutral, disagree, strongly disagree
Staining of RPD is absent | one year
  5-point Likert scale: strongly agree, agree, neutral, disagree, strongly disagree
Color stability is maintained | one year
  5-point Likert scale: strongly agree, agree, neutral, disagree, strongly disagree
Anatomic form of RPD is maintained | one year
  5-point Likert scale: strongly agree, agree, neutral, disagree, strongly disagree
Incidence of mechanical complications | one year
  Loosening or fracture of prosthetic components Nominal: O: absence; 1: presence
Incidence of biological complications | one year
  Presence of periodontal pathology Nominal: O: absence; 1: presence
Plaque accumulation around RPD abutment teeth. | one year
  Simplified Oral Hygiene Index (Greene and Vermelion, 1964). Ordinal: 0: no debris or stain present; 1: Soft debris covering not more than one third of the tooth surface, or presence of extrinsic stains without other debris regardless of surface area covered; 2: Soft debris covering more than one third, but not more than two thirds, of the exposed tooth surface; 3: Soft debris covering more than two thirds of the exposed tooth surface.
Bleeding around RPO abutment teeth | one year
  Gingival index (Loe and Silness 1963)'. Ordinal: 0: absence of inflammation/normal gingiva; 1: mild inflammation, slight change in color, slight edema, no bleeding on probing; 2: moderate inflammation, moderate glazing, redness, edema and hypertrophy, bleeding on probing; 3: severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
Probing pocket depths around RPD Dependent variable abutment teeth measured in millimeters | one year
  Measured through probing with a periodontal probe, evaluated on all tooth aspects. Scale: Distance between mucosal margin and probe stop measured in millimeters.
Mobility of RPO abutment teeth | one year
  Mobility classification (Miller 1950). Ordinal: 0: no detected mobility; 1: first sign of movement greater than normal; 2: up to 1 mm in any direction; 3: more than 1 mm in any direction and/or vertical depression.
ln mouth comfort | one year
  Visual analogue scale (0-10 cm); 0:very poor; 10: very good
Oral Health Impact Profile OHIP-14 | one year
  Oral Health Impact Profile OHIP-14 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Principal Investigator — Director of Research, Development and Education
Locations (1):
- Malo Clinic, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Anonymized database containing the study variables
Supporting Information: SAP
Time Frame: Upon study completion and for 8 years.
Access Criteria: Upon solicitation to the Investigators